CLINICAL TRIAL: NCT03608007
Title: Phase II, Open-Label, Single Arm Study of the Efficacy and Safety of X-396 Capsule in Patients With ROS1 Positive Advanced NSCLC
Brief Title: X-396 Capsule in Advanced NSCLC Patients With ROS1 Gene Rearrangement
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTP-42723
Record Dates: First submitted 2018-05-16; First posted 2018-07-31 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Lung Cancer; ROS1 Gene Rearrangement
Keywords: ROS1 NSCLC; X-396
MeSH Terms: conditions — Lung Neoplasms | interventions — ensartinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- X-396 Capsule (Experimental): Single-arm trial whereby all consented, enrolled, eligible patients receive X-396 capsule, 225 mg once daily.
  Interventions: Drug: X-396 Capsule

INTERVENTIONS:
Drug: X-396 Capsule — 225 mg once daily
  Other Names: Ensartinib

SUMMARY:
To assess treatment effectiveness and safety of oral X-396 capsule (Ensartinib) administered to Chinese patients with Advanced Non-Small Cell Lung Cancer (NSCLC) that is confirmed to be positive for a c-ROS Oncogene (ROS1) positive gene mutation (translocation or inversion).

DETAILED DESCRIPTION:
This is a phase II, multicenter, single-arm study in which the efficacy and safety of X-396 capsule (Ensartinib) will be assessed in adult Chinese patients with ROS1-positive (rearrangement or inversion) non-small cell lung cancer (NSCLC). Approximately 69 patients (59 for never-treated, and 10 for previously treated with crizotinib) with locally advanced or metastatic NSCLC carrying ROS1-rearrangement will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, 18 years of age or older
* Histologically or cytologically proven diagnosis of NSCLC that is locally advanced or metastatic
* Positive for translocation or inversion events involving the ROS1 gene
* Tyrosine kinase inhibitor (TKI) treatment-naive or have previously received no more than one systemic treatment regimen(s) such as chemotherapy (After a 3-week washout period)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Predicted survival ≥ 3 months
* Drug related toxicities were relieved to grade 1, except for hair loss (based on NCI CTCAE v4.03)
* Adequate organ function
* At least 1 measurable tumor lesion as per RECIST v1.1
* Asymptomatic central nervous system (CNS) metastases do not require the use of steroids or anticonvulsants.
* Signed and dated informed consent
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Agree to use effective contraception during the study period and for at least 90 days after completion of the study treatment

Exclusion Criteria:

* Current treatment on another systemic anti-cancer therapy
* Prior therapy specifically directed against ROS1 fusion genes (except for the exploratory arm that will enroll patients pretreated with crizotinib)
* Evidence of active malignancy within last 3 years
* Previous therapeutic clinical trial must have completed at least 4 week prior to initiation of study drug
* Prior surgery or immunotherapy must have completed at least 4 weeks, and radiation must have been completed at least 2 weeks prior to initiation of study drug
* Known interstitial fibrosis or interstitial lung disease
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of study medication
* Clinically significant cardiovascular disease
* Patients with a known allergy or delayed hypersensitivity reaction to study drug or its excipient
* Pregnant or breast feeding
* Use of drugs or foods that are known potent CYP3A4 inhibitors or inducers
* Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol
* Other serious illness or medical condition potentially interfering with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) based on independent radiology review (IRC) according to RECIST 1.1 | 12 weeks
  ORR per RECIST 1.1 calculated as the proportion of patients with a best overall response defined as complete response (CR) or partial response (PR), based on IRC.

SECONDARY OUTCOMES:
ORR based on investigator assessment according to RECIST 1.1 | 12 weeks
  ORR per RECIST 1.1 calculated as the proportion of patients with a best overall response defined as CR or PR, based on investigator's assessment
Disease control rate (DCR) according to RECIST 1.1 | 12 weeks
  DCR defined as the percentage of patients who have achieved CR, PR and stable disease (SD), based on RECIST 1.1 measured by IRC or investigator
Intracranial overall response rate (iORR) by IRC and investigator assessment according to RECIST 1.1 | 12 weeks
  iORR calculated as the ORR (CR+PR) of lesions in the brain for patients who have measurable disease in the brain at baseline.
Progression-free survival (PFS) based on IRC or investigator according to RECIST 1.1 | 36 months
  PFS defined as time from first dose of X-396 capsule to disease progression or death due to any cause, based on RECIST 1.1.
Time to progression (TTP) based on IRC or investigator according to RECIST 1.1 | 36 months
  TTP defined as time from first dose of X-396 capsule to disease progression, based on RECIST 1.1.
Duration of response (DOR) based on IRC or investigator according to RECIST 1.1 | 36 months
  DOR defined as time from documentation of tumor response (CR or PR) to disease progression or death, based on RECIST 1.1
Overall survival (OS) | 36 months
  OS, defined as time from first dose of X-396 to death due to any cause.
Change From Baseline Scores on the functional assessment of cancer therapy - Lung (FACT-L) quality of life questionnaire | 36 months
  The FACT-L questionnaire consisted of several major aspects of life (Physical, social/family, emotional, and functional well-being) as well as lung cancer subscale (symptoms, cognitive function, regret of smoking). Scores for item ranging from 0 (not at all) to 4 (very much).
Incidence of patients experiencing adverse events (AE) | 36 months
  Adverse events are graded according to CTCAE 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Principal Investigator — PHD
Locations (1):
- Chest hospital affiliated to Shanghai jiao tong university, Shanghai, Shanghai Municipality, China